CLINICAL TRIAL: NCT04825223
Title: Safety and Immunogenicity of an Investigational Multicomponent Meningococcal Group B Vaccine in Adults, Adolescents, Toddlers, and Infants
Brief Title: Study of a Novel Multicomponent Meningococcal Group B Vaccine When Given Alone or With Other Licensed Vaccines in Adults, Adolescents, Toddlers and Infants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision. Termination decision not related to any safety concern.
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAN00002; U1111-1244-0377 (Registry Identifier: ICTRP); 2023-506970-11 (Registry Identifier: CTIS); 2021-003070-31 (EudraCT Number)
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Meningococcal Immunisation; Healthy Volunteers
MeSH Terms: interventions — MenB-FHbp vaccine; 4CMenB vaccine; DNA, Recombinant; DNA, Ribosomal; Elements

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 4 stages, sequentially:
  * Stage 1: adults and adolescents from the US, equally randomized to 8 vaccine groups
  * Stage 2; adults and adolescents from the EU and the US, equally randomized to 11 vaccine groups
  * Stage 3: toddlers from the EU, equally randomized to 6 vaccine groups
  * Stage 4: infants from the EU, equally randomized to 6 vaccine groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage 1 and Stage 2 (adults and adolescents) will be modified double-blind: the investigators and study staff who conduct the safety assessment and the participant will not know which vaccine is administered. Only the study staff who prepare and administer the vaccine and are not involved with the safety evaluation will know which vaccine is administered. The individual(s) responsible for the preparation / administration of the vaccines will not be authorized to collect any safety or serology data. Testing laboratories will be blinded. In order to maintain the blind in Stage 2 (adults and adolescents), a placebo injection will be used. After the 6-months safety assessment from the last dose of primary vaccination, Stage 2 will be unblinded for the administration of booster vaccinations. Stage 3 and Stage 4 (toddlers and infants) will be open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Stage 1: MenB vaccine formulation(s) (Experimental): Assigned MenB vaccine formulation or Placebo single injection in the respective dosing schedule at Day 01, Day 31 and Day 181
  Interventions: Drug: Meningococcal Group B Vaccine MenB; Drug: Placebo
- Stage 1: vaccine comparator(s) (Active Comparator): Bexsero vaccine or Trumenba vaccine or Placebo single injection in the respective dosing schedule at Day 01, Day 31 and Day 181
  Interventions: Drug: Multicomponent Meningococcal B Vaccine; Drug: Meningococcal Group B Vaccine (recombinant deoxyribonucleic acid [rDNA], component, adsorbed); Drug: Placebo
- Stage 2: MenB vaccine formulation(s) (Experimental): Assigned MenB vaccine formulation, MenQuadfi vaccine and Placebo single injection in the respective dosing schedule at Day 01, Day 31, Day 61 and Day 181 + booster dose of leading MenB vaccine formulation single injection at Day 366
  Interventions: Drug: Meningococcal Group B Vaccine MenB; Drug: Placebo; Drug: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine MenACYW conjugate vaccine
- Stage 2: vaccine comparator(s) (Active Comparator): Bexsero vaccine or Trumenba vaccine and Placebo single injection in the respective dosing schedule at Day 01, Day 31, Day 61 and Day 181 + booster dose of Bexsero vaccine single injection at Day 366
  Interventions: Drug: Multicomponent Meningococcal B Vaccine; Drug: Meningococcal Group B Vaccine (recombinant deoxyribonucleic acid [rDNA], component, adsorbed); Drug: Placebo
- Stage 3: Men B vaccine formulation(s) (Experimental): Assigned MenB vaccine formulation and/or MenQuadfi vaccine single injection in the respective dosing schedule at Day 01 and Day 61
  Interventions: Drug: Meningococcal Group B Vaccine MenB; Drug: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine MenACYW conjugate vaccine
- Stage 3: MenQuadfi vaccine and vaccine comparator (Active Comparator): MenQuadfi vaccine single injection at Day 01 or Bexsero vaccine single injection at Day 01 and Day 61
  Interventions: Drug: Meningococcal Group B Vaccine (recombinant deoxyribonucleic acid [rDNA], component, adsorbed); Drug: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine MenACYW conjugate vaccine
- Stage 4: MenB vaccine formulation(s) (Experimental): Assigned MenB vaccine formulation, Routine Vaccines (RV)s and MenQuadfi vaccine single injection in the respective dosing at 2 months of ages [moa] (Day 01), 4moa (Day 61) and 12 moa
  Interventions: Drug: Meningococcal Group B Vaccine MenB; Drug: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine MenACYW conjugate vaccine
- Stage 4: MenQuadfi vaccine and vaccine comparator (Active Comparator): MenQuadfi vaccine or Bexsero vaccine and RVs in the respective dosing schedule at 2 months of ages [moa] (Day 01), 4moa (Day 61) and 12 moa
  Interventions: Drug: Meningococcal Group B Vaccine (recombinant deoxyribonucleic acid [rDNA], component, adsorbed); Drug: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine MenACYW conjugate vaccine

INTERVENTIONS:
Drug: Multicomponent Meningococcal B Vaccine — Pharmaceutical form:Liquid suspension for injection in a single vial Four liquid suspensions and one diluent (only for Stage 1) Route of administration: Intramuscular
  Other Names: Trumenba®
  Arms: Stage 1: vaccine comparator(s); Stage 2: vaccine comparator(s)
Drug: Meningococcal Group B Vaccine MenB — Pharmaceutical form:Liquid suspension for injection in a pre-filled syringe Route of administration: Intramuscular
  Other Names: MenB
  Arms: Stage 1: MenB vaccine formulation(s); Stage 2: MenB vaccine formulation(s); Stage 3: Men B vaccine formulation(s); Stage 4: MenB vaccine formulation(s)
Drug: Meningococcal Group B Vaccine (recombinant deoxyribonucleic acid [rDNA], component, adsorbed) — Pharmaceutical form:Liquid suspension for injection in a pre-filled syringe Route of administration: Intramuscular
  Other Names: Bexsero®
  Arms: Stage 1: vaccine comparator(s); Stage 2: vaccine comparator(s); Stage 3: MenQuadfi vaccine and vaccine comparator; Stage 4: MenQuadfi vaccine and vaccine comparator
Drug: Placebo — Pharmaceutical form:Liquid solution for injection in a vial Route of administration: Intramuscular
  Arms: Stage 1: MenB vaccine formulation(s); Stage 1: vaccine comparator(s); Stage 2: MenB vaccine formulation(s); Stage 2: vaccine comparator(s)
Drug: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine MenACYW conjugate vaccine — Pharmaceutical form:Liquid solution for injection in a vial Route of administration: Intramuscular
  Other Names: MenQuadfi™
  Arms: Stage 2: MenB vaccine formulation(s); Stage 3: Men B vaccine formulation(s); Stage 3: MenQuadfi vaccine and vaccine comparator; Stage 4: MenB vaccine formulation(s); Stage 4: MenQuadfi vaccine and vaccine comparator

SUMMARY:
Primary Objective:

* To describe the safety profile of the SP MenB vaccine formulations and the 2 licensed MenB comparator vaccines in healthy adults, adolescents, toddlers and infants, when administered alone (Stages 1-4) or concomitantly with MenQuadfiTM (MenACYW conjugate vaccine) (for Stages 2-4 only), and with age-appropriated routine pediatric vaccines (for Stages 3-4 only)

  1. To describe the safety profile of the SP MenB vaccine formulations, Bexsero Vaccine and Trumenba Vaccine in healthy adults, and adolescents;
  2. To describe the safety profile of the SP MenB vaccine formulations and Bexsero Vaccine in toddlers and infants;
  3. To describe the safety profile of the SP MenB vaccine formulations,

     * when administered alone
     * when administered with MenQuadfiTM (MenACYW conjugate vaccine)
     * when administered with routine infant immunizations
* To describe the immune response to the SP MenB vaccine formulations and the 2 licensed MenB comparator vaccines after the last dose of primary vaccination in healthy adults, adolescents, toddlers and infants, when administered alone, or concomitantly with MenQuadfi Vaccine or other routine vaccines, as measured by the serum bactericidal assay using human complement (hSBA) in the primary panel of MenB strains by Stage, by age group and by vaccine schedule

Secondary Objective:

* To describe the immune response to the SP MenB vaccine formulations and the 2 licensed MenB comparator vaccines at each timepoint in healthy adults, adolescents, toddlers and infants, when administered alone or concomitantly with MenQuadfi Vaccine or other routine vaccines as measured by hSBA in the primary panel of MenB strains by Stage by age group and by vaccine schedule
* To describe the immune response (breadth of coverage) in the secondary panel of MenB strains in participants (adults and adolescents) in Stage 1 and 2 after the last dose of the primary series in each group
* To describe the persistence of immune response following primary series at D366, and immune response 1 month after a booster dose of the SP MenB vaccine given 1-year post-dose 1 (at D366) in a subset of adults and adolescents in Stage 2 who received SP MenB vaccine formulations, Bexsero Vaccine or Trumenba Vaccine as measured by hSBA in the primary panel of MenB strains by age group
* To describe the immune response against meningococcal serogroups A, C, W and Y measured with hSBA in participants from each agegroup receiving MenQuadfi Vaccine

DETAILED DESCRIPTION:
Study duration per participant will be approximately: 7 months for Stage 1 participants, 12 to 18.5 months for Stage 2 participants, 12 months for Stage 3 participants and 18 months for Stage 4 participants

In each vaccine group at each age group (Stage 1, 3 and 4 only), the first 5 participants enrolled (sentinels) will be assessed via early safety data review (ESDR) as a cohort for the evaluation of biological safety and overall safety profile for D01-D08 post dose 1. The safety data collected will be reviewed before proceeding with recruitment of remaining participants in each study group. Enrollment of remaining participants randomized to each group will be based on the outcome of the safety assessments of the sentinels: only a positive review outcome will allow the enrollment of the sentinel cohort of the respective lower age group.

ELIGIBILITY:
Inclusion criteria :

-For US: Aged 10 to 25 years on the day of inclusion ("10-25 years" means from the day of the 10th birthday to the day before the 26th birthday) For EU: Aged 42 to 89 days or 12 to 18 months or 10 to 50 years on the day of inclusion ("42 to 89 days" means from 42 days after birth to the 89th day after birth; "12-18 months" means from the12th month after birth to the day before the 19th month after birth; "10-50 years" means from the day of the 10th birthday to the day before the 51st birthday Participants or participant and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures Covered by health insurance (applicable depending on local regulations) Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and judgement of the Investigator

For adults: A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

* Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile OR
* Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to the first study intervention administration until at least 4 weeks after the last study intervention administration.

A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) the day of any dose of study intervention

For adolescents: A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

* Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be pre-menarche OR
* Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to the first study intervention administration until at least 4 weeks after the last study intervention administration A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) the day of any dose of study intervention -For infants: Born at full term of pregnancy (≥37 weeks) and with a birth weight ≥2.5 kg or born after a gestation period of 27 through 36 weeks and medically stable as assessed by the investigator, based on the following definition: "Medically stable" refers to the condition of premature infants who do not require significant medical support or ongoing management for debilitating disease and who have demonstrated a clinical course of sustained recovery by the time they receive the first dose of study intervention - - -

Exclusion criteria:

-Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months or since birth for infants and toddlers; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months or since birth for infants and toddlers) History of any Neisseria meningitidis infection, confirmed either clinically, serologically, or microbiologically At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease) Individuals with active tuberculosis Known systemic hypersensitivity to latex or to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances For adults and adolescents: Self-report of thrombocytopenia, contraindicating intra-muscular (IM) vaccination * For infants and toddlers: Laboratory-confirmed thrombocytopenia, or known thrombocytopenia, as reported by the parent/legally acceptable representative contraindicating intramuscular vaccination Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination For infants and toddlers: History of intussusception Receipt of any vaccine in the 4 weeks (28 days) preceding the first trial vaccination or planned receipt of any vaccine 4 weeks before to 4 weeks after each trial vaccination or study visit with collection of blood for immunogenicity assessments, except for influenza vaccination, which may be received at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines Previous vaccination against meningococcal B disease with either the study vaccines or another licensed or investigational vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroup B) For infants and toddlers: Previous vaccination against meningococcal disease with either the study vaccines or any other licensed or investigational vaccine containing serogroups A, C, W, Y; or meningococcal serogroup B Receipt of immune globulins, blood or blood-derived products in the past 3 months or since birth for infants and toddlers Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first immunogenicity blood draw For infants: Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, hepatitis A, measles, mumps, rubella, varicella; and Haemophilus influenzae type b, Streptococcus pneumoniae, and /or rotavirus infection or disease, and receipt of more than 1 previous dose of hepatitis B vaccine Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion Moderate or severe acute illness/infection (according to the investigator's judgment), febrile illness (temperature ≥ 38.0°C or ≥ 100.4°F). A prospective participant should not be enrolled in the study until the condition has resolved or the febrile event has subsided History of Guillain-Barré syndrome History of any neurologic disorders, including any seizures and progressive neurologic disorders Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily For adults and adolescents: Identified as an investigator or employee of the investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the investigator or employee with direct involvement in the proposed study For infants and toddlers: Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study For adults and adolescents: Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 42 Days to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 576 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events (AEs) | Within 30 minutes after vaccination
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Number of participants with solicited injection site reactions or systemic reactions | Within 7 days after vaccination
  Adverse reactions pre-listed in the protocol and case report form (CRF) Injection site reactions: pain, erythema and swelling (or tenderness, erythema and swelling for infants and toddlers) Systemic reactions: fever, headache, malaise, myalgia (or fever, vomiting, crying abnormal, drowsiness, appetite lost, irritability for infants and toddlers)
Number of participants with unsolicited AEs | Within 30 days after vaccination
  AEs that do not fulfill the conditions of solicited reactions
Number of participants with serious adverse events (SAEs) | Up to 6 months after last vaccination
  SAEs reported throughout the study, including adverse events of special interest (AESI)s
Number of participants with medically attended adverse events (MAAE)s | Up to 6 months after last vaccination
  AEs with a new onset or a worsening of a condition that prompts the participant or participant's parent/guardian to seek unplanned medical advice at a physician's office or Emergency Department
Number of participants with out-of-range biological test results | From baseline (pre-vaccination) up to Day 07 (post-vaccination)
  Out-of-range biological test results occurring in the sentinel cohorts of each age group
Antibody titers in the primary panel of MenB strains before primary vaccination | Day 01 (pre-vaccination)
  Antibody titers measured by serum bactericidal assay using human complement (hSBA)
Antibody titers in the primary panel of MenB strains after primary vaccination | Day 30 (post-vaccination)
  Antibody titers measured by hSBA

SECONDARY OUTCOMES:
Antibody titers in the primary panel of MenB strains after each vaccination | Day 01, Day 31, Day 61, Day 91, Day 181, Day 211, Day 366 and Day 396
  Antibody titers measured by hSBA
Antibody titers in the secondary panel of MenB strains (stage 1 and 2 only) | Day 01 (pre-vaccination) and Day 30 (post-vaccination)
  Antibody titers measured by hSBA
Antibody titers in the primary panel of MenB strains (stage 2 only) | Day 366 (pre-vaccination) and Day 396 (post-vaccination)
  Antibody titers measured by hSBA
Antibody titers against each of Men A, C, W, and Y strains | Day 01 (pre-vaccination) and Day 30 (post-vaccination)
  Antibody titers measured by hSBA in participants receiving MenQuadfi vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- United States (8):
  - Lakeview Clinical Research Site Number : 8400029, Guntersville, Alabama
  - California Research Foundation Site Number : 8400005, San Diego, California
  - PAS Research Site Number : 8400032, Tampa, Florida
  - Brengle Family Medicine Site Number : 8400044, Indianapolis, Indiana
  - AMR El Dorado Site Number : 8400018, El Dorado, Kansas
  - Alliance for Multispecialty Research LLC Site Number : 8400013, Wichita, Kansas
  - Prime Global Research, Inc. Site Number : 8400043, The Bronx, New York
  - The Research Center of the Upstate Site Number : 8400008, Greenville, South Carolina
- Puerto Rico (2):
  - Investigational Site Number : 6300003, Ponce
  - Investigational Site Number : 6300001, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAN00002 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25368&tenant=MT_SNY_9011